CLINICAL TRIAL: NCT05226338
Title: A Phase 1, Open-Label, Randomized, Single Dose, 3-Period, 3-Treatment Study to Evaluate the Relative Bioavailability of D-0502 Tablet Formulations in Healthy Female Subjects
Brief Title: Evaluation of Relative Bioavailability of D-0502 Tablet in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D0502-104
Record Dates: First submitted 2021-10-22; First posted 2022-02-07 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Healthy Female Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): 3 period, 3 dose level
  Interventions: Drug: D-0502
- Sequence 2 (Experimental): 3 period, 3 dose level
  Interventions: Drug: D-0502
- Sequence 3 (Experimental): 3 period, 3 dose level
  Interventions: Drug: D-0502
- Sequence 4 (Experimental): 3 period, 3 dose level
  Interventions: Drug: D-0502
- Sequence 5 (Experimental): 3 period, 3 dose level
  Interventions: Drug: D-0502
- Sequence 6 (Experimental): 3 period, 3 dose level
  Interventions: Drug: D-0502

INTERVENTIONS:
Drug: D-0502 — Formulation 1 Formulation 2 Formulation 3

SUMMARY:
Relative Bioavailability study of D-0502 tablet formulation in healthy female subjects

DETAILED DESCRIPTION:
Phase 1, Open Label, Randomized, Single dose, 3 Period, 3 treatment study to evaluation the relative Bioavailability of D-0502 tablet formulation in healthy female subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects between the ages of 18-55
* Required evaluation by Investigator for screening and enrollment
* Agreement and compliance with the study and follow-up procedures

Exclusion Criteria:

* Significant medical history or current comorbidly determined by the Investigator.
* Pregnant or nursing women

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Access the oral bioavailability of D-0502 100mg and 200mg tablets | Single Dose, 3 period, 3 treatment study separated by 14 day washout periods to evaluate safety and bioavailability. Overall time in study is approximately 42 days.
  Access the oral bioavailability of D-0502 100mg and 200mg tablets relative to D-0502 50mg tablet formulation

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No